CLINICAL TRIAL: NCT07102407
Title: Effect of a Constructivist Educational Program on Preventing Ventilator-Associated Pneumonia in Intensive Care Units
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Karaman Training and Research Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 05- 2024/05
Record Dates: First submitted 2025-07-28; First posted 2025-08-03 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-06

CONDITIONS: Ventilator Associated Pneumonia
MeSH Terms: conditions — Pneumonia, Ventilator-Associated

STUDY DESIGN:
Intervention Model Description: An interventional study with a one-month intervention period and a six-month post-intervention period follow-up.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- ICU with trained staff (Experimental): The intensive care unit where nurses and cleaning staff will receive a routine VAP prevention program and constructive training
  Interventions: Other: Contructivist; Other: Routine training
- ICU with non-trained staff (Experimental): The Intensive care unit, where nurses and cleaning staff will receive only routine training for the prevention of VAP
  Interventions: Other: Routine training

INTERVENTIONS:
Other: Contructivist — Implementation of constructivist training on VAP in small groups
  Other Names: Constructivist Educational Program about VAP
  Arms: ICU with trained staff
Other: Routine training — Implementation of routine training on VAP in large groups
  Other Names: Routine training about preventing VAP

SUMMARY:
This study is designed to investigate the impact of a constructivist education program on nurses and cleaning personnel regarding the preventive care bundle for the prevention of ventilator-associated pneumonia in the intensive care unit.

DETAILED DESCRIPTION:
Ventilator-associated pneumonia (VAP) is one of the types of healthcare-associated infections seen in critically ill patients receiving mechanical ventilation. VAP is defined as a nosocomial lower respiratory tract infection that begins 48 hours or more after the initiation of invasive mechanical ventilation in intubated patients. VAP leads to increased mortality and morbidity, prolonged hospital stay, and economic and psychological costs. Prevention of VAP has primarily been achieved through the "package approach," which involves the simultaneous implementation of various preventive strategies for all patients. Therefore, it is important to conduct educational programs for healthcare personnel to reduce the incidence of VAP. Learning in constructivist education is based on establishing connections between existing and new knowledge and integrating each new piece of information into existing knowledge. While constructivist education and routine training are provided to the staff of one of the two adult intensive care units included in this study, only routine training is offered to the staff of the other. VAP data in intensive care units with constructivist education and routine training will be compared. Constructivist education will be provided to intensive care nursing and cleaning staff in small groups and over a total period of one month. The data from both intensive care units will be examined comparatively within six months after the completion of the constructivist training.

After the implementation of the constructivist education, all patients in the ICU will be included in the study.

ELIGIBILITY:
Inclusion Criteria:

* age > 18 years
* patients receiving mechanical ventilation for more than 48 hours

Exclusion Criteria:

* A clinical diagnosis of pneumonia at the time of admission

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Estimated)
Dates: Start 2025-08-15 (Actual); Primary Completion 2026-02-15 (Estimated); Study Completion 2026-02-18 (Estimated)

PRIMARY OUTCOMES:
prevalence of VAP among patients ( the number of patients diagnosed with VAP during the study period | 6 months period
  The prevalence of VAP will be compared between two intensive care units over a 6-month period after implementing an educational program for nurses and cleaning staff on the preventive care bundle for VAP prevention.

CONTACTS AND LOCATIONS:
Overall Officials: Saliha Yarımoglu, MD, Principal Investigator — Karaman Training and Research Hospital
Locations (1):
- Karaman Training and Research Hospital, Karaman, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No